CLINICAL TRIAL: NCT00284635
Title: Fast-Track vs Conventional for UKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: KF-01-231/03
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2007-07-04 (Estimated); Status verified 2007-07

CONDITIONS: Unicompartmental Knee Replacement

INTERVENTIONS:
Procedure: Fast track vs conventional

SUMMARY:
The purpose of this study is to see if it is possible to discharge patient undergoing a UKA 1 day postoperatively

ELIGIBILITY:
Inclusion Criteria:

* UKA, ASA I-II

Exclusion Criteria:

* medical history of abdominal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: arne borgwardt, M.D., Principal Investigator — Frederiksberg University Hospital
Locations (1):
- Frederiksberg University Hospital, Copenhagen, Frederiksberg C, Denmark